CLINICAL TRIAL: NCT02339636
Title: A Clinical Study of Subclinical Enthesitis and Synovitis in Patients With Vulgaris Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The 306 Hospital of People's Liberation Army (Other)
Responsible Party: Sponsor
Other Study IDs: 306PLA-002
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2013-08

CONDITIONS: Vulgaris Psoriasis
Keywords: subclinical, enthesitis, synovitis
MeSH Terms: conditions — Synovitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case group: 100 patients with vulgaris psoriasi without arthritis
  Interventions: Other: PDUS examination
- control group: 100 age-matched patients with other skin diseases without arthritis
  Interventions: Other: PDUS examination

INTERVENTIONS:
Other: PDUS examination

SUMMARY:
A clinical study of subclinical enthesitis and synovitis in patients with vulgaris psoriasis

DETAILED DESCRIPTION:
A total of 100 patients with vulgaris psoriasis and 100 age-matched controls with other skin diseases, all without musculoskeletal diseases, will be recruited. They will undergo dermatological assessment and a blinded PDUS evaluation. Clinical assessment included demographics, severity of psoriasis, musculoskeletal clinical examination and sport activities. PDUS evaluation consisted of the detection of grey scale (GS) synovitis and synovial PD signal in joints of extremities, GS enthesopathy and entheseal PD signal in entheses of lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* age≥18years
* patients with vulgaris psoriasis(dur
* patients with other skin diseases without musculoskeletal disorders
* no joint involvement and no clinical symptoms and signs of enthesitis and synovitis

Exclusion Criteria:

* BMI≥24
* have history of gout or arthritis or peripheral neurological disease of lower extremity or trauma
* have received any systemic therapy(i.e.NSAIDs, corticosteroids, immunosuppressants, retinoids or biological agents) in 3 months
* pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both patients with psoriasis and patients with other skin diseases
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of subclinical enthesitis and synovitis | one and a half year
  To investigate the incidence of subclinical enthesitis and synovitis in patients with vulgaris

SECONDARY OUTCOMES:
Number of participants with Risk factors of subclinical enthesitis and synovitis | one and a half year
  To find out predictor factors of subclinical enthesitis and synovitis in patients with vulgaris psoriasis

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Liu, M.D., Principal Investigator — The 306 Hospital of People's Liberation Army
Locations (1):
- 306 Hospital of PLA, Beijing, China